CLINICAL TRIAL: NCT03681340
Title: Investigation of the Caries Prevention and Remineralization Effects of Hydroxyapatite Toothpaste
Brief Title: Remineralization Effects of Hydroxyapatite Toothpaste
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Joachim Enax (Industry)
Responsible Party: Sponsor-Investigator, Dr. Joachim Enax, Senior Scientist, Dr. Kurt Wolff GmbH & Co. KG
Organization: Dr. Kurt Wolff GmbH & Co. KG (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REHT18
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Caries, Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxyapatite toothpaste (Experimental): 4 weeks toothbrushing with a hydroxyapatite toothpaste
  Interventions: Other: Hydroxyapatite toothpaste; Other: Fluoridated toothpaste
- Fluoridated toothpaste (Active Comparator): 4 weeks toothbrushing with a fluoridated toothpaste
  Interventions: Other: Hydroxyapatite toothpaste; Other: Fluoridated toothpaste

INTERVENTIONS:
Other: Hydroxyapatite toothpaste — If in a subject a significant increase of carious lesions will be observed, her/his parents are informed about the necessity for further caries preventive measures (e.g. dietary changes, use of fluoride products, reduction of cariogenic microflora with chlorhexidine, xylitol chewing gum, etc.) and caries preventive treatment (removing caries and placing a restoration) by the study centers is offered.
Other: Fluoridated toothpaste — If in a subject a significant increase of carious lesions will be observed, her/his parents are informed about the necessity for further caries preventive measures (e.g. dietary changes, use of fluoride products, reduction of cariogenic microflora with chlorhexidine, xylitol chewing gum, etc.) and caries preventive treatment (removing caries and placing a restoration) by the study centers is offered.

SUMMARY:
The objective of this in situ clinical study is to determine whether a toothpaste containing hydroxyapatite microclusters is as effective as a fluoridated kid's toothpaste in promoting remineralization of early caries lesions and inhibiting the development of caries lesions.

DETAILED DESCRIPTION:
The investigators hypothesize that (1) both the hydroxyapatite and the fluoridated toothpaste promote caries remineralization that is significantly greater than zero, and (2) the two toothpaste formulations are equally effective with respect to post-treatment remineralization and inhibition of demineralization.

* Non-inferiority will be considered established if there is no statistically significant difference in percentage of remineralization between the hydroxyapatite-containing toothpaste and the fluoridated kid's toothpaste for any one measurement method.
* Superiority/inferiority will be considered established if at least 20% statistically significant difference is observed between the hydroxyapatite-containing toothpaste and the fluoridated kid's toothpaste for any one measurement method

ELIGIBILITY:
Inclusion Criteria:

1. Male and/or female subjects 18 to 50 years inclusive
2. Minimum of 20 natural uncrowned teeth (excluding third molars) must be present
3. Willing to wear retainer 24 hours per day
4. No active, unrestored cavities
5. Have normal salivary flow rate (stimulated and unstimulated flow of ≥0.7 ml/min and ≥0.2 ml/min respectively) ascertained from a preliminary sialometry test
6. Available throughout entire study
7. Willing to use only assigned products for oral hygiene throughout the duration of the study
8. Must give written informed consent
9. Must be in good general health
10. No known history of allergy to personal care/consumer products or their ingredients, relevant to any ingredient in the test products as determined by the dental/medical professional monitoring the study

Exclusion Criteria:

1. Advanced periodontal disease
2. Medical condition which requires premedication prior to dental visits/procedures
3. Not enough teeth to secure the oral retainer
4. Diseases of the soft or hard oral tissues
5. Wearing of an orthodontic retainer(s)
6. Impaired salivary function
7. Current use of drugs that can affect salivary flow
8. Use of antibiotics one (1) month prior to or during this study
9. Positive urine test for pregnancy or self-reported breastfeeding. A urine pregnancy test will be performed on female subjects of child-bearing potential.
10. Participation in another clinical study one (1) week prior to the start of the washout period or during this study period
11. Use of tobacco products
12. Allergic history to common toothpaste ingredients
13. Allergic history to amino acids
14. Immune compromised individuals (HIV, AIDS, immuno-suppressive drug therapy) as determined by review of medical history

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Caries remineralization | 4 weeks
  Analyis of mineral gain/loss and lesion depth by microradiography

CONTACTS AND LOCATIONS:
Overall Officials: Bennett T. Amaechi, Prof., Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amaechi BT, AbdulAzees PA, Alshareif DO, Shehata MA, Lima PPCS, Abdollahi A, Kalkhorani PS, Evans V. Comparative efficacy of a hydroxyapatite and a fluoride toothpaste for prevention and remineralization of dental caries in children. BDJ Open. 2019 Dec 9;5:18. doi: 10.1038/s41405-019-0026-8. eCollection 2019. PMID 31839988